CLINICAL TRIAL: NCT02862756
Title: Analysis of Thrombo-embolic Complications After Endovascular Treatment of Unruptured Intracranial Aneurysms
Acronym: ACET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR16021*
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-03

CONDITIONS: Unruptured Intracranial Aneurysms
MeSH Terms: interventions — Restraint, Physical

ARMS (1):
- patient with endovascular treatment (Experimental)
  Interventions: Other: diffusion-weighted MRI and clinical examination

INTERVENTIONS:
Other: diffusion-weighted MRI and clinical examination

SUMMARY:
Endovascular treatment of ruptured and unruptured intracranial aneurysms presents complications, mainly the thrombo-embolic complication. No specific studies have been conducted to study factors associated with the occurrence of thromboembolic complications (symptomatic or not) post endovascular treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
In this multicenter, prospective study, patients with treatment of unruptured intracranial aneurysms will be recruited. The thromboembolic complications will be research using diffusion-weighted MRI.

ELIGIBILITY:
Inclusion Criteria:

* patient having a programmed endovascular treatment for unruptured intracranial aneurysm
* patient older than 18 years
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program

Exclusion Criteria:

* patients with contraindications for MRI
* patients whose clinical condition does not allow sufficient cooperation to the realization of MRI
* patients with arteriovenous malformation intracranial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Thromboembolic complication | 72 hours after endovascular treatment
  Thromboembolic complication diagnosed using diffusion-weighted MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Derived] Pierot L, Rouchaud A, Chabert E, Desal H, Ricolfi F, Barbe C, Soize S, Zerroug A, Eugene F, Clarencon F, Ferre JC. Endovascular treatment of unruptured intracranial aneurysms: Rate of thromboembolic events depicted by diffusion-weighted imaging in relation to different techniques. J Neurointerv Surg. 2025 Aug 13;17(9):949-955. doi: 10.1136/jnis-2024-022051. PMID 39095086